CLINICAL TRIAL: NCT01437111
Title: A Phase III (Phase IV Program) Open-Label, Multicenter Clinical Trial in Thailand to Study the Effect of MK-217A/Alendronate Sodium 70-mg/Vitamin D3 5600 IU Combination Tablet (Fosamax Plus 70/5600) for 6 Months on 25-Hydroxyvitamin D Levels in the Treatment of Osteoporosis in Postmenopausal Women and Men
Brief Title: Study of MK-217A/Alendronate Sodium 70-mg/Vitamin D3 5600 IU Combination Tablet (MK-0217A-329)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0217A-329
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Cholecalciferol; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fosamax Plus (Experimental): Calcium supplement (elemental calcium and/or calcium carbonate) without vitamin D will also be supplied to participants
  Interventions: Drug: MK-217A/Alendronate Sodium 70-mg/Vitamin D3 5600 IU Combination Tablet

INTERVENTIONS:
Drug: MK-217A/Alendronate Sodium 70-mg/Vitamin D3 5600 IU Combination Tablet — One combination tablet orally once a week
  Other Names: Fosamax Plus 70/5600

SUMMARY:
This study will assess the effect of 26 weeks of once-weekly treatment with MK-217A/Alendronate Sodium 70-mg/Vitamin D3 5600 IU Combination Tablet (Fosamax Plus 70/5600) on serum levels of 25-hydroxyvitamin D [25(OH)D].

ELIGIBILITY:
Inclusion Criteria:

* Man aged 50 or older, or a woman who is postmenopausal on day of signing informed consent or has been menopausal for at least one year
* Meets bone mineral density (BMD) criteria
* Agree to discontinue any osteoporosis drug treatment for duration of study

Exclusion Criteria:

* Any contraindication to alendronate and vitamin D
* Not ambulatory
* Has received treatment with any anabolic steroid agent within the past 12 months, systemic glucocorticoids, for more than 2 weeks in the past 6 months, current use of immunosuppressants, fluoride treatment at a dose greater than 1 mg/day for more than 2 weeks within the past 3 months, treated with parathyroid hormone (PTH) for more than 2 weeks within the past 3 months, current use of chemotherapy or heparin, use of growth hormone for more than 2 weeks within the past 6 months, use of active hormonal vitamin D analogs in the past 2 months, current use of vitamin A >10,000 IU daily, current use of, lithium, or anti-convulsants including barbiturates, hydantoins, and carbamazepine, current use of calcium supplement in amount excess of 1500 mg daily, and/or current use of Vitamin D supplement
* History of malignancy <5 years, except adequately treated basal cell or squamous cell skin cancer and in situ cervical cancer
* One or more of the following concomitant conditions: Upper gastrointestinal (GI) disorders not adequately controlled; myocardial infarction, unstable angina, stroke and revascularization condition within 3 months; malabsorption syndrome; primary or secondary hyperparathyroidism not adequately treated; thyroid disease not adequately controlled; severe renal insufficiency; uncontrolled genitourinary, cardiovascular, hepatic, renal, endocrine, hematologic, neurological, psychiatric, or pulmonary diseases; uncontrolled hypertension; new onset diabetes (within 3 months), poorly controlled hyperglycemia, or hypoglycemia for any cause; evidence for metabolic bone disease other than osteoporosis; abnormal indices of calcium metabolism; and/or active renal stone disease
* User of illicit recreational drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence
* Heavy consumer of alcohol or alcohol containing products.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-10-26 (Actual); Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Songpatanasilp T, Rojanasthien S, Sugkraroek P, Ongphiphadhanakul B, Robert L, Robert CS, Luevitoonvechkij S, Santora AC. Open-label study of treatment with alendronate sodium plus vitamin D in men and women with osteoporosis in Thailand. BMC Musculoskelet Disord. 2018 Nov 6;19(1):392. doi: 10.1186/s12891-018-2309-y. PMID 30400864

RESULTS

PARTICIPANT FLOW:
Groups:
- Fosamax Plus: All Participants: All participants who were enrolled in the study to receive one oral combination tablet of Fosamax Plus weekly.
Period: Overall Study
Arm/Group | Fosamax Plus: All Participants
Started | 200
Treated Participants | 198
Completed | 182
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Not reported | 5
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis was performed on the All Patients as Treated (APaT) population, which included all participants who received treatment. Of 200 participants enrolled in the study, baseline data were not provided for two participants who did not receive treatment.
Groups:
- Fosamax Plus: All Treated Participants: All participants who received at least one oral dose combination tablet of Fosamax Plus.
Arm/Group | Fosamax Plus: All Treated Participants
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age data were not reported for 2 participants.
  Years | 68.81 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data were not reported for 2 participants.
  Participants
    Female | 193
    Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serum 25-hydroxyvitamin D >=50 ng/mL at Week 26
Description: Serum samples to measure serum 25-hydroxyvitamin D [25(OH)D] will be collected at specific visits during the treatment phase of the study.
Time Frame: Week 26
Population: Full Analysis Set (FAS) consisted of participants who received >=1 dose of study drug; had >=1 post-baseline observation for the analysis endpoint; and had baseline data. For analysis, participants in the FAS were categorized into 3 subgroups by osteoporosis therapy received at baseline: Recent/Current, Other therapy, and Treatment Naïve
Measure: Number; unit: Participants
Groups:
- Fosamax Plus: Recent/Current Osteoporosis Therapy at Baseline: Participants receiving recent/current osteoporosis therapy at baseline (including bisphosphonate, strontium, estrogen, or SERM were administered open-label alendronate sodium 70 mg+Vitamin D3 5600 IU combination tablet (Fosamax Plus D) orally once a week for 26 weeks.
- Fosamax Plus: Other Osteoporosis Therapy at Baseline: Participants receiving other osteoporosis drugs at baseline (besides bisphosphonate, strontium, estrogen, or SERM) were administered open-label alendronate sodium 70 mg+Vitamin D3 5600 IU combination tablet (Fosamax Plus D) orally once a week for 26 weeks.
- Fosamax Plus: Treatment Naive at Baseline: Participants that were treatment-naïve or not recently treated at baseline were administered open-label alendronate sodium 70 mg+Vitamin D3 5600 IU combination tablet (Fosamax Plus D) orally once a week for 26 weeks.
Arm/Group | Fosamax Plus: Recent/Current Osteoporosis Therapy at Baseline | Fosamax Plus: Other Osteoporosis Therapy at Baseline | Fosamax Plus: Treatment Naive at Baseline | Fosamax Plus: All Treated Participants
Number analyzed (Participants) | 28 | 64 | 94 | 186
Participants | 1 | 3 | 1 | 5

2. Secondary Outcome: Mean Percent Change From Baseline of Bone Resorption Marker of Serum Beta-CrossLaps at Week 26
Description: Serum samples for Beta-CrossLaps (β-CTx) will be collected at specific visits during the treatment phase of the study.
Time Frame: Baseline and Week 26
Population: Per Protocol Population consisted of FAS but excluded participants who had important deviations from protocol or did not complete study on study drug. For analysis, participants in Per Protocol Population were categorized into 3 subgroups by osteoporosis therapy received at baseline: Recent/Current, Other therapy, and Treatment Naïve.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Fosamax Plus: Recent/Current Osteoporosis Therapy at Baseline | Fosamax Plus: Other Osteoporosis Therapy at Baseline | Fosamax Plus: Treatment Naive at Baseline | Fosamax Plus: All Treated Participants
Number analyzed (Participants) | 28 | 62 | 92 | 182
Percent change | -12.65 (56.94) | -49.82 (35.08) | -76.81 (20.33) | -57.74 (40.34)

ADVERSE EVENTS:
Time Frame: Up to Week 26
Description: Of 200 participants enrolled in the study, two participants did not receive treatment and were not evaluated for safety.
Arm/Group | Fosamax Plus: All Treated Participants
Serious Adverse Events (participants affected / at risk) | 4/198
Other Adverse Events (participants affected / at risk) | 10/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosamax Plus: All Treated Participants (N=198)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Tongue neoplasm, malignant stage, unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosamax Plus: All Treated Participants (N=198)
Upper respiratory tract infection (Infections and infestations) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to allow the Sponsor to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Investigators have also agreed that any information identified by the SPONSOR as confidential must be deleted prior to submission.